CLINICAL TRIAL: NCT03594201
Title: A Retrospective Study on the Effect of Male Progressive Sperm Count After Semen Pretreatment on ICSI Fertilization Outcome
Status: Completed | Type: Observational
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Responsible Party: Sponsor
Other Study IDs: KYXM-201803
Record Dates: First submitted 2018-07-11; First posted 2018-07-20 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2018-07

CONDITIONS: Sperm Count, Low; Reproductive Sterility
Keywords: ICSI, progressive sperm count, embryo
MeSH Terms: conditions — Oligospermia; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- group1: A+B grade sperm count after treatment=0
  Interventions: Other: semen pretreatment
- group2: 0<A+B grade sperm count after treatment≤10^6
  Interventions: Other: semen pretreatment
- group3: 10^6<A+B grade sperm count after treatment<2*10^6
  Interventions: Other: semen pretreatment
- group4: A+B grade sperm count after treatment≥2*10^6
  Interventions: Other: semen pretreatment

INTERVENTIONS:
Other: semen pretreatment — semen pretreatment

SUMMARY:
The investigators plan to retrospectively analyze clinical data from 14,189 fresh ICSI cycles in Reproductive and Genetic Hospital of CITIC-Xiangya from January 2016 to December 2017.The investigators will regard total progressive sperm number of 2 x 10^6 after pretreatment as the boundary value, and will divide total progressive sperm number of 2 x 10^6 after pretreatment into 2 x 10^6 or higher and < 2 x 10^6 groups, and will further divide < 2 x 10^6 group into: = 0, (0,10^6], (10^6, 2 x 10^6) three groups. Propensity score matching will be used to balance the baseline data between four groups. The matching variables are age, female BMI, AFC, AMH and ICSI.

ELIGIBILITY:
Inclusion Criteria:

* infertility female and sterility male for reproductive treatment

Exclusion Criteria:

* chromosomal abnormalities
* none retrieval oocyte
* none oocyte for ICSI
* Recurrent abortion
* female age≥37 years
* Assisted hatching
* abnormal oocyte zona pellucida
* In Vitro Maturation
* AZF microdeletion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infertile couples take ART treament due to poor male semen quality.
Sampling Method: Non-Probability Sample
Enrollment: 12215 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-03 (Actual)

PRIMARY OUTCOMES:
high quality embryo rate for ICSI | two years
  rate of embryo grade above 6CI on the third day after fertilization

SECONDARY OUTCOMES:
fertilization rate of ICSI | two years
  number of fertilized oocytes/ number of metaphase II oocytes
normal fertilization rate of ICSI | two years
  number of 2PN fertilized oocytes/ number of metaphase II oocytes

CONTACTS AND LOCATIONS:
Overall Officials: Liang Hu, MD,PHD, Principal Investigator — Reproductive & Genetic Hospital of CITIC-Xiangya
Locations (1):
- Reproductive & Genetic Hospital of CITIC-XIANGYA, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No